CLINICAL TRIAL: NCT03045029
Title: ADAPT - A Patient Registry of the Real-world Use of Orenitram®
Acronym: ADAPT
Status: Active, not recruiting | Type: Observational
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TDE-PH-401
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Oral Treprostiinil; Orenitram
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 78 Weeks
Biospecimen Retention: Samples With DNA — 1. Optional evaluation of biomarkers
  2. Optional evaluation of pharmacogenomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oral treprostinil: Sustained-release oral tablets for three times daily (TID) administration in prostacyclin naive and prostacyclin transition patients
  Interventions: Drug: Oral treprostinil

INTERVENTIONS:
Drug: Oral treprostinil — Sustained-release oral tablets for TID administration
  Other Names: Treprostinil diethanolamine; Treprostinil diolamine

SUMMARY:
This prospective, observational, multicenter, patient registry will follow patients who are receiving treatment with Orenitram for the treatment of PAH for up to 78 weeks from Orenitram initiation

ELIGIBILITY:
INCLUSION CRITERIA

Patients are eligible for the registry if:

1. The patient voluntarily gives informed consent to participate in the study.
2. The patient must be at least 18 years of age or older.
3. The patient is prescribed Orenitram (per the package insert indication), and plans to initiate therapy with this medication or has been receiving Orenitram for 182 or fewer days.
4. The patient agrees to dosing, prostacyclin-related AE of interest record keeping, survey participation during designated time periods, and recording any medication changes, use, for the duration of the study.
5. The patient has the ability to answer surveys and use the diary in English.
6. The patient must have an email address and be willing to access the PRO Portal.

EXCLUSION CRITERIA

Patients are ineligible for the registry if:

1. The patient has previously received Orenitram for more than 182 days.
2. The patient is currently participating in an investigational drug or device study or has participated in a clinical study with an investigational product other than Orenitram in PAH within

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible if they have been receiving Orenitram for 182 or fewer days.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Real-world use and tolerability of Orenitram in new starts and prostacyclin transition patients | Baseline to Week 78

SECONDARY OUTCOMES:
To assess treatment-related outcomes during routine clinical care. | Baseline to Week 78
  eg, 6-Minute Walk Distance [6MWD], World Health Organization [WHO] Functional Class [FC]
To observe the development, timing, severity, frequency, and treatment of prostacyclin-related adverse events (AEs) of interest | Baseline to Week 78
Use of concomitant medications | Baseline to Week 78
To evaluate information on clinical titration schedules implemented for transition to and from alternative prostacyclin-class therapies | Baseline to Week 78
Healthcare resource utilization trends | Baseline to Week 78
Health-related quality of life in PAH and treatment satisfaction | Baseline to Week 78
To evaluate reasons for discontinuation of Orenitram | Baseline to Week 78
To evaluate titration and dosing schedules of Orenitram | Baseline to Week 78

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - University of California - San Francisco, Fresno, California
  - University of Southern California - Keck Medical Center, Los Angeles, California
  - Paloma Medical Group, San Juan Capistrano, California
  - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - Harbor UCLA Medical Center, Torrance, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Pueblo Pulmonary Associates, Pueblo, Colorado
  - Lung Associates PA, Bradenton, Florida
  - University of Florida Clinical Research Center, Gainesville, Florida
  - St. Vincent's Lung, Sleep, and Critical Care Specialists, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - USF South Florida Heart Health, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Healthcare/Research, Austell, Georgia
  - Loyola University Chicago, Chicago, Illinois
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University Of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville Physicians Outpatient Center, Louisville, Kentucky
  - Chest Medicine Associates, South Portland, Maine
  - Mclaren Greater Lansing, Okemos, Michigan
  - Beaumont Hospital Troy, Troy, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Pulmonary Health Physicians, PC, Fayetteville, New York
  - Stony Brook University Medical Center, Islandia, New York
  - Northwell Health- Long Island Jewish Forest Hills, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Pinehurst Medical Clinic, INC., Pinehurst, North Carolina
  - Lima Memorial Hospital, Lima, Ohio
  - INTEGRIS Nazih Zuhdi Transplant Institution, Oklahoma City, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pittsburgh - Heart and Vascular Medicine Institute, Pittsburgh, Pennsylvania
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - Center for Biomedical Research, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Heart Care Associates, LLC, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No